CLINICAL TRIAL: NCT02490969
Title: Copeptin Registry (proCORE) Biomarkers in Cardiology (BIC)-19
Acronym: proCORE
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Martin Moeckel, Univ. Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: BIC 19
Record Dates: First submitted 2015-06-25; First posted 2015-07-07 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Acute Myocardial Infarction
Keywords: copeptin; rule out marker, emergency department, cheast pain unit; emergency department; chest pain unit
MeSH Terms: conditions — Diabetes Insipidus; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Routine management observation — Early rule out of myocardial infarction with combined copetine and troponin testing at admission

SUMMARY:
Registry of an interventional Study-proved Strategy (BIC-8) using Copeptin and Troponin for the Early Rule-Out of Acute Myocardial Infarction (AMI) in Patients with Suspected Acute Coronary Syndrome (ACS) and a low-to intermediate risk profile.

DETAILED DESCRIPTION:
Registry of an interventional Study-proved Strategy (BIC-8) using Copeptin and Troponin for the Early Rule-Out of Acute Myocardial Infarction (AMI) in Patients with Suspected Acute Coronary Syndrome (ACS) and a low-to intermediate risk profile.

Primary objective:

To monitor the safety of the early rule-out strategy using combined testing of copeptin and troponin at admission of patients with signs and symptoms suggestive of ACS and a low- to intermediate risk profile, who are discharged or moved to another hospital after testing copeptin and troponin negative (defined as copeptin below 10 pmol/l and cardiac troponin below 99th percentile URL).

Secondary objectives:

* To monitor routine application of the early rule-out strategy, patient characteristics, risk profile of all patients tested for copeptin and troponin at admission, irrespective of their biomarker test result
* To monitor diagnoses, clinical course and outcome of all patients tested for copeptin and troponin at admission

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Emergency Department or CPU with signs and symptoms consistent with acute coronary syndrome
* Low-to intermediate risk profile (GRACE-score below 140 and a low- to intermediate likelihood of ACS as judged by the treating physician)
* Patients eligible for the early rule-out strategy using combined copeptin and troponin testing at admission, irrespective of biomarker test results and disposition decision
* full-aged patient

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women who present to an ED/CPU with signs and symptoms suggestive of acute coronary syndrome (NSTE-ACS) and an intermediate-to low risk profile in whom an early rule-out strategy for AMI is applied and who therefore undergo single combined troponin and copeptin testing at admission as part of standard management.
Sampling Method: Non-Probability Sample
Enrollment: 2256 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  One-month all-cause mortality in patients in whom acute myocardial infarction is ruled-out using the early rule-out strategy and who are therefore discharged from the ED

CONTACTS AND LOCATIONS:
Overall Officials: Martin Moeckel, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on reasonable request

REFERENCES:
- [Derived] Giannitsis E, Clifford P, Slagman A, Ruedelstein R, Liebetrau C, Hamm C, Honnart D, Huber K, Vollert JO, Simonelli C, Schroder M, Wiemer JC, Mueller-Hennessen M, Schroer H, Kastner K, Mockel M. Multicentre cross-sectional observational registry to monitor the safety of early discharge after rule-out of acute myocardial infarction by copeptin and troponin: the Pro-Core registry. BMJ Open. 2019 Jul 23;9(7):e028311. doi: 10.1136/bmjopen-2018-028311. PMID 31340965